CLINICAL TRIAL: NCT07047144
Title: A Phase 2, Double-Blind Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy, and Safety of Apitegromab in Subjects <2 Years Old With Spinal Muscular Atrophy (SMA)
Brief Title: A Study to Evaluate How Apitegromab Works in Subjects Who Are Less Than 2 Years Old and Have Spinal Muscular Atrophy
Acronym: OPAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRK-015-005
Expanded Access: NCT06877689 (Available)
Record Dates: First submitted 2025-04-16; First posted 2025-07-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Spinal Muscular Atrophy; SMA; Spinal Muscular Atrophy Type 2; Spinal Muscular Atrophy Type 3; Neuromuscular Manifestations; Anti-myostatin
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Neuromuscular Manifestations | interventions — apitegromab; nusinersen; Risdiplam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor, the subject's caregiver, Investigators, and site personnel, with the exception of the designated unblinded personnel (eg, site Pharmacist), will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apitegromab low dose + SMN Therapy (Experimental): Patients who are less than 2 years of age with SMA will receive apitegromab every 4 weeks by intravenous (IV) infusion during the 48-week Treatment Period.
  Patients must have been treated with an approved SMN1-targeted therapy (ie, onasemnogene abeparvovec-xioi) or are continuing to be treated with an approved SMN2-targeted therapy (ie, nusinersen or risdiplam).
  Interventions: Drug: Apitegromab; Drug: Nusinersen; Drug: Risdiplam
- Apitegromab high dose + SMN Therapy (Experimental): Patients who are less than 2 years of age with SMA will receive apitegromab every 4 weeks by intravenous (IV) infusion during the 48-week Treatment Period.
  Patients must have been treated with an approved SMN1-targeted therapy (ie, onasemnogene abeparvovec-xioi) or are continuing to be treated with an approved SMN2-targeted therapy (ie, nusinersen or risdiplam).
  Interventions: Drug: Apitegromab; Drug: Nusinersen; Drug: Risdiplam

INTERVENTIONS:
Drug: Apitegromab — Apitegromab is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that specifically binds to human pro/latent myostatin with high affinity inhibiting myostatin activation. SRK-015 will be administered every 4 weeks by intravenous (IV) infusion.
  Other Names: SRK-015
Drug: Nusinersen — Nusinersen is a current standard-of-care SMN therapy that targets the SMN2 gene. It will be administered intrathecally per the prescribing information.
  Other Names: Spinraza
Drug: Risdiplam — Risdiplam is a current standard-of-care SMN therapy that targets the SMN2 gene. It will be administered orally per the prescribing information.
  Other Names: Evrysdi

SUMMARY:
This double-blind, Phase 2, multiple-dose study will be conducted to evaluate the PK/PD, efficacy, safety, and tolerability of apitegromab in subjects <2 years old with 5q autosomal recessive SMA who have delayed motor milestones for their age attributed to SMA at the discretion of the Investigator or a Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) score <55.

ELIGIBILITY:
Inclusion Criteria:

1. Is <2 years old at the time of the informed consent
2. Had a gestational age of ≥35 weeks and gestational body weight ≥2.0 kg at birth
3. Has confirmed diagnosis of 5q autosomal recessive SMA
4. Has confirmed presence of SMN2 gene copy(ies)
5. Must have been treated with an approved SMN1-targeted therapy (ie, onasemnogene abeparvovec-xioi) or are continuing to be treated with an approved SMN2-targeted therapy (ie, nusinersen or risdiplam)
6. Body weight for age is no less than 1st percentile based on the WHO Child Growth Standards at the Screening Visit
7. Has delayed motor milestones for age attributed to SMA at the discretion of the Investigator or a CHOP-INTEND score <55

Exclusion Criteria:

1. Nutritional status that is not anticipated to be stable throughout the study or medical necessity for a gastric feeding tube, where most feeds are administered by this route
2. Major orthopedic issues such as severe scoliosis or severe contractures or interventional procedure, including spine or hip surgery, which is considered to have the potential to substantially limit the ability of the subject to be evaluated on any motor function outcome measures, within 6 months before Screening or anticipated during the study
3. Any other physical limitations (eg, the subject requires cast for contractures) that would prevent the subject from undergoing motor function outcome measures throughout the study.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the PK of apitegromab in subjects <2 years old with SMA | 52 Weeks
  Apitegromab concentrations in serum
Evaluate the PD of apitegromab in subjects <2 years old with SMA | 52 Weeks
  Total latent myostatin concentrations in serum
Evaluate the motor function outcomes (ie, efficacy) due to apitegromab treatment | 48 Weeks
  Change from baseline in the raw score of the Bayley Scale of Infant and Toddler Development, Fourth Edition - Gross Motor Subscale (BSID-4 GMS) at 48 weeks. BSID-4 GMS is a standardized assessment commonly used to evaluate development across 5 domains in infants and young children. It consists of 58 items, scored from 0 to 2 for each item, with higher scores indicating better gross motor development.

SECONDARY OUTCOMES:
Assess the safety and tolerability of apitegromab administered to subjects receiving an SMN therapy | 52 Weeks
  Incidence of TEAEs and SAEs by severity

CONTACTS AND LOCATIONS:
Locations (14):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford Neuroscience Health Center (SNHC), Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Neurology Rare Disease Center, Flower Mound, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
- Belgium (2):
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHR Citadelle, Liège
- Italy (2):
  - Fondazione I.R.C.C.S. - Istituto Neurologico Carlo Besta, Milan
  - Centro Clinico NeMO Milano - Fondazione Serena Onlus, Milan
- Spain (2):
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Universitari i Politecnico La Fecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No